CLINICAL TRIAL: NCT05751941
Title: A Phase II Randomized Study of Sipuleucel-T With or Without Continuing New Hormonal Agents (NHA) in Metastatic Prostate Cancer With PSA Progression While on NHA and LHRH Analog
Brief Title: Study of Sipuleucel-T With or Without Continuing New Hormonal Agents in Metastatic Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-22003
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Metastatic Prostate Cancer
Keywords: PSA Progression
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone; enzalutamide; apalutamide; sipuleucel-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sipuleucel-T with NHA (Experimental): Participants will continue taking New Hormonal Agents (NHA) while receiving sipuleucel-t as standard of care.
  Interventions: Drug: Abiraterone; Drug: Enzalutamide; Drug: Apalutamide; Drug: Sipuleucel-T
- Sipuleucel-T without NHA (Experimental): Participants will discontinue use of New Hormonal Agents (NHA) while receiving sipuleucel-t as standard of care.
  Interventions: Drug: Sipuleucel-T

INTERVENTIONS:
Drug: Abiraterone — 1000 mg of Abiraterone will be given orally daily plus prednisone 5-10 mg daily
  Arms: Sipuleucel-T with NHA
Drug: Enzalutamide — 160 mg of Enzalutamide will be given orally daily ending at week 4
  Other Names: Xtandi
  Arms: Sipuleucel-T with NHA
Drug: Apalutamide — 240 mg of Apalutamide will be given orally daily ending at week 4
  Arms: Sipuleucel-T with NHA
Drug: Sipuleucel-T — Sipuleucel-T is considered standard of care and will be infused into the participant three times at approximately 2-week intervals starting week 0, 2 and 4.
  Other Names: Provenge

SUMMARY:
This study is designed to test the hypothesis that using Sipuleucel-T (Provenge) in combination with new hormonal agents (NHA) (abiraterone, enzalutamide, apalutamide) for the treatment of participants with asymptomatic metastatic castration resistant prostate cancer (mCRPC) and no visceral metastases would enhance the activation of antigen presenting cells (APC) by sipuleucel-T.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic or minimally symptomatic metastatic prostate cancer, and the diagnosis of prostate cancer needs to be histologically confirmed by biopsy of the prostate or a metastatic lesion
* On combined ADT with LHRH analog and a NHA (enzalutamide, apalutamide or abiraterone) for metastatic prostate cancer with PSA progression, but no imaging progression based on the prostate cancer working group (PCWG) 3 criteria
* Age 18 or above
* ECOG performance status 0 or 1
* Participants must have adequate organ and marrow function as defined below:
* Absolute neutrophil count ≥1,000/mcL
* Platelets ≥100,000/mcL
* Hemoglobin > 10 g/dl
* AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
* Creatinine 1.5 ≤ institutional ULN
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of sipuleucel-T are eligible for this trial
* No uncontrolled arrhythmia: patients with h/o myocardial infarction or history of congestive heart failure, need to have estimated left ventricle ejection fraction above 40% either on echocardiogram or MUGA scan within 6 months of study enrollment
* Non-sterilized men who are sexually active with a female partner of childbearing potential must agree to use adequate contraception prior to the study enrollment, and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study
* Prior treatment with sipuleucel-T
* Participants who have not recovered from adverse events (AEs) due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 2).
* Participants who require > 50% dose reduction of NHA are excluded from the study except for taking abiraterone at 250 mg with low fat food
* Documented brain metastases or liver metastases
* Treatment with any investigational compound within 30 days prior to the first dose of Sipuleucel-T
* Documented brain metastases or liver metastases
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome. HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for sipluleucel-T to be less clinically active in this population
* Inability to comply with protocol requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative APC Activation | At Week 4
  Cumulative APC activation is calculated as the sum of APC activation across 0, 2, and 4 weeks

SECONDARY OUTCOMES:
Time to PSA progression | Up to week 44
  PSA progression will be defined as the time from randomization to the first date of documented PSA progression based on the prostate cancer working group (PCWG) 3 criteria.
Radiographic Progression Free Survival | Up to week 44
  Radiographic Progression Free Survival (rPFS) as assessed by conventional CT and bone scan
IgG Responses | At week 14
  To evaluate increases in IgG levels after treatment, pre- and post treatment signal intensities from Luminex xMAP will be compared using a one-sided paired Wilcoxon signed-rank test. To evaluate whether the fold changes in IgG levels after treatment were higher in the NHA group than the without NHA group, the values from the two groups will be compared using a one-sided Wilcoxon rank-sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Jingsong Zhang, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided